CLINICAL TRIAL: NCT05162781
Title: Transferring Speed of Processing Gains to Everyday Cognitive Tasks After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Posit Science (Unknown)
Responsible Party: Principal Investigator, Gitendra Uswatte, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300008211; 1R01AG070049-01A1 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2021-12-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Cognitive Dysfunction
Keywords: stroke; cognitive dysfunction; cognitive processing speed; IADL
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Half of the participants will receive CICT, which consists of SOPT, IADL training in the lab, and a Transfer Package targeting IADL performance outside it. The other half will receive BF-HELP, which consists of SOPT, in-lab training on relaxation, nutrition, and sleep hygiene, and a Transfer Package targeting implementation of these lifestyle changes outside it. Half of the CICT group will receive 9 follow-up phone calls over the course of six months. The other CICT participants will receive none. The same will apply to the BF-HELP group. The phone calls will support integration of the behavioral changes targeted during treatment to everyday life afterwards.
  For all participants, outcome testing will take place one month before treatment (Baseline 1), one day before treatment (Baseline 2 aka Pre-treatment), one day afterwards (Post-treatment), and 6-months afterwards (6-month Follow-up). Randomization will take place after Baseline 2.
Who Masked: Outcomes Assessor
Masking Description: Tester will be blinded to group assignment of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CICT with Follow-up Phone Calls (Experimental): Participants in this group will receive 35 hours of training. Ten 1-hour sessions of SOPT will be scheduled in the home with training conducted independently by participants. Ten 2.5 hours of in-lab, face-to-face, therapist directed sessions will be scheduled. These sessions will feature a brief period of SOPT; the bulk of the sessions will be committed to (A) shaping on IADL and (B) the Cognitive Transfer Package. Training sessions will be permitted to be scheduled over 2-4 weeks. Family caregivers will receive training on how to best support participants in their therapeutic program. After treatment ends, four phone calls will be placed once-a-week for four weeks, then once-a-month for 5 months. The follow-up calls will target transition of any changes achieved during treatment into everyday life on a long-term basis.
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Instrumental Activities of Daily Living In-lab Training; Behavioral: Cognitive Transfer Packagke; Behavioral: Family Caregiver Coaching; Behavioral: Follow-up Phone Calls
- CICT without Follow-up Phone Calls (Experimental): Participants in this group will receive 35 hours of training. Ten 1-hour sessions of SOPT will be scheduled in the home with training conducted independently by participants. Ten 2.5 hours of in-lab, face-to-face, therapist directed sessions will be scheduled. These sessions will feature a brief period of SOPT; the bulk of the sessions will be committed to (A) shaping on IADL and (B) the Cognitive Transfer Package. Training sessions will be permitted to be scheduled over 2-4 weeks. Family caregivers will receive training on how to best support participants in their therapeutic program. No follow-up phone calls will be made after treatment ends.
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Instrumental Activities of Daily Living In-lab Training; Behavioral: Cognitive Transfer Packagke; Behavioral: Family Caregiver Coaching
- BF-HELP with Follow-up Phone Calls (Active Comparator): Participants in this group will receive 35 hours of training. Ten 1-hour sessions of SOPT will be scheduled in the home with training conducted independently by participants. Ten 2.5 hours of in-lab, face-to-face, therapist directed sessions will be scheduled. These sessions will feature a brief period of SOPT; the bulk of the sessions will be committed to (A) training on relaxation, healthy nutrition, and healthy sleep, and (B) the Healthy Lifestyle Transfer Package. Training sessions will be permitted to be scheduled over 2-4 weeks. Family caregivers will receive training on how to best support participants in their therapeutic program. After treatment ends, four phone calls will be placed once-a-week for four weeks, then once-a-month for 5 months. The follow-up calls will target transition of any changes achieved during treatment into everyday life on a long-term basis.
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Family Caregiver Coaching; Behavioral: Follow-up Phone Calls; Behavioral: Healthy Lifestyle In-lab Training; Behavioral: Healthy Lifestyle Transfer Package
- BF-HELP without Follow-up Phone Calls (Active Comparator): Participants in this group will receive 35 hours of training. Ten 1-hour sessions of SOPT will be scheduled in the home with training conducted independently by participants. Ten 2.5 hours of in-lab, face-to-face, therapist directed sessions will be scheduled. These sessions will feature a brief period of SOPT; the bulk of the sessions will be committed to (A) training on relaxation, healthy nutrition, and healthy sleep, and (B) the Healthy Lifestyle Transfer Package. Training sessions will be permitted to be scheduled over 2-4 weeks. Family caregivers will receive training on how to best support participants in their therapeutic program. No follow-up phone calls will be made after treatment ends.
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Family Caregiver Coaching; Behavioral: Follow-up Phone Calls; Behavioral: Healthy Lifestyle In-lab Training; Behavioral: Healthy Lifestyle Transfer Package

INTERVENTIONS:
Behavioral: Speed of Processing Training — This training component targets cognitive processing speed, i.e., how quickly individuals process information that they receive through their senses. Cognitive processing speed is thought to be a basic capacity of the brain that underlies several other cognitive functions. Training is implemented using a web-based computer "game", in which participants are required to fixate on a target at the center of the screen and identify targets in the periphery. The game is made progressively more difficult, in small increments, as participants gain mastery by increasing the speed at which targets are presented and increasing the number of distractors.
  Other Names: SOPT
Behavioral: Instrumental Activities of Daily Living In-lab Training — The training component is thought to bridge SOPT training, which targets a basic cognitive capacity, and IADL performance in daily life. This training component will involve repeated trials in which participants will practice carrying out simulated IADL tasks in the lab under the supervision of the trainer. The training will follow shaping principles, i.e., task requirements will be made progressively more challenging, in small increments, as participants gain mastery. Frequent, positive feedback will be provided.
  Other Names: IADL In-lab Training
  Arms: CICT with Follow-up Phone Calls; CICT without Follow-up Phone Calls
Behavioral: Cognitive Transfer Packagke — This training component is designed to transfer improvements in cognition from the treatment setting to everyday life. Elements of this package include negotiating a behavioral contract about the roles of the participant and family caregiver in the treatment, monitoring behavior outside the lab, and assigning performance of IADL as homework.
  Arms: CICT with Follow-up Phone Calls; CICT without Follow-up Phone Calls
Behavioral: Family Caregiver Coaching — One or more family members of the participant will receive coaching on how to best support the participant in carrying out the in-home components of the intervention.
Behavioral: Follow-up Phone Calls — After treatment ends, four phone calls will be placed once-a-week for four weeks, then once-a-month for 5 months. The follow-up calls will target transition of any changes achieved during treatment into everyday life on a long-term basis after.
  Arms: BF-HELP with Follow-up Phone Calls; BF-HELP without Follow-up Phone Calls; CICT with Follow-up Phone Calls
Behavioral: Healthy Lifestyle In-lab Training — This training component is designed to promote lifestyle changes that support brain fitness. Participants will receive education and coaching in the lab on relaxation, healthy nutrition, and healthy sleep.
  Arms: BF-HELP with Follow-up Phone Calls; BF-HELP without Follow-up Phone Calls
Behavioral: Healthy Lifestyle Transfer Package — This training component is designed to support integration into everyday life of the lifestyle changes training in the lab. Elements of this package include negotiating a behavioral contract about the roles of the participant and family caregiver in the treatment, monitoring behavior outside the lab, and assigning relaxation exercises, for example, as homework.
  Arms: BF-HELP with Follow-up Phone Calls; BF-HELP without Follow-up Phone Calls

SUMMARY:
This study will compare two approaches to cognitive rehabilitation in adults with stroke with persistent, mild to moderate, cognitive impairment. Both approaches will feature a web-based computer "game" that trains cognitive processing speed, i.e., how quickly individuals process information that they receive through their senses. This training is termed Speed of Processing Training (SOPT). One approach will add (A) in-lab training on everyday activities with important cognitive components and (B) procedures designed to transfer improvements in cognition from the treatment setting to everyday life. This approach is termed Constraint-Induced Cognitive Therapy (CICT). The other approach will add (A) in-lab training on relaxation, healthy nutrition, and healthy sleep and (B) procedures designed to promote integration of these lifestyle changes into everyday life. This approach is termed Brain Fitness-Heath Education Lifestyle Program (BF-HELP).

Both CICT and BF-HELP will involve 35 hours of training. Ten 1-hour sessions of SOPT will be scheduled in the home with training conducted independently by participants. Ten 2.5 hours of in-lab, face-to-face, therapist directed sessions will be scheduled. These sessions will feature a brief period of SOPT; the bulk of the sessions will be committed to in-lab training on the target behaviors and the procedures designed to promote transfer of therapeutic gains to daily life; The set of the latter procedures is termed the Transfer Package. To accommodate the demands of participants' other activities, training sessions will be permitted to be scheduled as tightly as every weekday over 2 weeks or as loosely as every other weekday or so over 4 weeks. Family caregivers in both groups will also receive training on how to best support participants in their therapeutic program.

The study will also test if there is an advantage to placing follow-up phone calls after treatment ends. The purpose of the calls will be to support transition of any behavioral changes achieved during treatment into everyday life on a long-term basis.

Participants will be randomly assigned to the interventions.

Testing will happen one month before treatment, one day before treatment, one day afterwards, and 6-months afterwards. Outcomes measured will include cognitive processing speed, cognitive function on laboratory tests, and spontaneous performance of everyday activities with important cognitive components in daily life.

ELIGIBILITY:
Primary Inclusion Criteria:

* stroke > 3 months previously
* mild-to-moderate general cognitive impairment as determined by a Montreal Cognitive Assessment (MOCA) score between 10-26
* some impairment in performance of daily activities; this will be determined by a score of 3.5 or below on the Cognitive Task Activity Log (CTAL)

Additional Inclusion Criteria:

* 40 years or older; no upper limit if medically stable
* sufficiently fit, from both a physical and mental health perspective, to take part in study
* adequate sight and hearing to complete UFOV test
* adequate thinking skills, e.g., ability to follow directions, retain information, to complete UFOV and CTAL, as marked by judgement of the screener that the candidate is able to adequately complete the UFOV and CTAL
* reside in the community (as opposed to a hospital or skilled nursing facility)
* able to travel to laboratory on multiple occasions
* caregiver available

Exclusion Criteria:

* cognitive impairment due to a developmental disability, psychiatric disorder, or substance abuse or due to another type of brain injury, such a traumatic brain injury, or a progressive brain disease, such as Alzheimer's Dementia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Neurological Disorders Measures (Neuro-QOL), Cognitive Function Scale | Change from Day 30 to Day 60, i.e., from Pre- to Post-treatment
  The Neuro-QOL assesses function in daily life in several domains; it is a widely used, validated, transdiagnostic, self-report measure. The development and use of the Neuro-QOL is supported by the National Institutes of Health. The component of the Neuro-QOL that assessed cognitive function will be used here. Items are rated by respondents using a five-point scale: 1 = not at all, 5 = very much. Higher scores indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Gitendra Uswatte, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States